CLINICAL TRIAL: NCT04795206
Title: A Retrospective Cohort Analysis of the Natural Disease Progression of Patients With Choroideremia in Real-World Clinical Practice
Brief Title: Natural Disease Progression in Participants With Choroideremia
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-CHM-11761
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Choroideremia
Keywords: X-linked inherited retinal disorder; Rare disease; Bilateral disease
MeSH Terms: conditions — Choroideremia; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Main Cohort: All eligible participants with CHM in IRIS Registry will be included.
  Interventions: Other: No Intervention
- Cohort 2: Trial-Matched Cohort: Only male participants with CHM from Cohort 1 to match Biogen's IST study population using propensity score matching will be included.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to quantify disease progression measured by best corrected visual acuity (BCVA) in the real-world setting among Choroideremia (CHM) participants. The secondary objectives are to describe demographic and baseline clinical characteristics among CHM participants and to match CHM participants in the Intelligent Research in Sight (IRIS®) Registry to Biogen's investigator sponsored trial (IST) study population using propensity score matching.

DETAILED DESCRIPTION:
This study is a retrospective cohort study of CHM eyes and participants which will include all eligible participants and eyes with the first documented diagnosis of CHM from July 1st, 2013 to December 31st, 2019 that meet the study criteria. This study will be conducted using data from American Academy of Ophthalmology's (AAO) IRIS® Registry which captures CHM participant's demographics, clinical characteristics and clinical outcomes from 2013.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1: All CHM Participants

* Participants with a documented diagnosis of CHM identified by the presence of International Classification of Diseases (ICD)-9/10 or SNOMED coding:

  1. ICD-9: 363.55
  2. ICD-10: H31.2
  3. SNOMED-CT: 75241009

Cohort 2: Trial-Matched CHM Participants

* Male participants with a documented diagnosis of CHM identified by the presence of ICD-9/10 or SNOMED coding:

  1. ICD-9: 363.55
  2. ICD-10: H31.21
  3. SNOMED-CT: 75241009

Key Exclusion Criteria:

* N/A

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Main cohort will include all eligible CHM participants in IRIS registry. Trial-matched cohort will include only male CHM participants from Cohort 1 to match Biogen's IST study population using propensity score matching.
Sampling Method: Non-Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Progression of Best Corrected Visual Acuity (BCVA) in Relation to Age | Up to 6 years
Percentage of Participants with Progression of BCVA Over Time After the Baseline BCVA | Up to 6 years

SECONDARY OUTCOMES:
Percentage of Participants with Demographics Described at Baseline | Up to 6 years
  The demographics will include age, sex, race, geographic region and treating provider specialty.
Matching Participants with CHM in the IRIS® Registry to Biogen's IST Study Population Using Propensity Score (PS) Matching | Up to 6 years
  A propensity score matching approach will be performed to select eligible male CHM participants from IRIS Registry to match Biogen's IST study population. With the approach, the probability of participating in the IST study given the observed baseline participant characteristics will be estimated for each participant. Propensity score will be estimated using logistic regression and pre-specified baseline covariates including participants demographics and clinical characteristics. The propensity match will be considered adequate if all the variables between the PS-matched CHM cohort and IST study cohort have an absolute value of the standardized mean difference (SMD) in PS-score that is less than 0.1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/